CLINICAL TRIAL: NCT01779063
Title: Promoting Adherence to Lymphedema Self-care in Breast Cancer Survivors
Brief Title: Promoting Adherence to Lymphedema Self-care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Sheila Ridner, Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 124137-RSG-13-022-01-CPPB
Record Dates: First submitted 2013-01-23; First posted 2013-01-30 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Lymphedema Self-care
Keywords: lymphedema; self-care; breast cancer
MeSH Terms: conditions — Lymphedema; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- web based multimedia intervention (Experimental): interactive,web based multimedia intervention
  Interventions: Behavioral: web based multimedia intervention
- education booklet (Active Comparator): printed educational booklet
  Interventions: Other: educational booklet

INTERVENTIONS:
Behavioral: web based multimedia intervention — cognitive therapy based web intervention
  Arms: web based multimedia intervention
Other: educational booklet — patient education booklet
  Arms: education booklet

SUMMARY:
Lymphedema is a chronic condition that causes physical and emotional challenges to breast cancer survivors. As a progressive condition, lymphedema can result in swelling/fibrosis that can impair function, promote infection, and cause discomfort and emotional distress. Daily self-care that is required to manage lymphedema is time-consuming, burdensome, and lifelong. Previous studies found that about half of breast cancer survivors with lymphedema do not complete self-care as directed. Feelings of being helpless to manage the condition, a desire to be normal, lack of noticeable results from self-care, and poor social/healthcare professional support are barriers to performing self-care on a regular basis. There is a need to develop and test interventions to promote effective self-care. Experts suggest the best self-care interventions should include patient perspectives and be available a readily accessible format. Technological advancements support use of innovative, creative approaches, such as Web-based multimedia interventions. Web-based interventions can be used in rural and urban settings. The investigators are proposing to develop a Web-based, multimedia intervention and a "take home" manual to support self-care in breast cancer survivors with lymphedema. The investigators plan to conduct focus groups with these survivors to determine the content and delivery format(s) and to help us identify breast cancer survivors with lymphedema for the video component. The investigators will then develop an intervention that will include self-care demonstrations and other supportive information to help patients to cope with the challenges of self-care. The focus groups will reconvene, review the intervention, and give us feedback on modifying and refining the intervention. After finalizing the intervention, The investigators will recruit more breast cancer survivors with lymphedema and provide one half of them an education booklet and the other half the Web-based intervention (or an alternative format such as DVD). Then, over 12 months, the investigators will periodically assess and compare both groups on self-care behaviors, physical and emotional concerns, and other issues such as money spent on lymphedema treatment. The group that receives the education booklet will be given access to the Web-based intervention after the 12 month follow-up is done, but the investigators will not ask them to complete any more forms.

This project builds upon the investigators prior work that has provided information about lymphedema self-care problems and the investigators previous experience in developing patient education videos and manuals. By providing accessible, detailed self-care instructions and a psychosocial component, this intervention has the potential to improve lymphedema self-care. If successful, this intervention can be offered to the larger national and international community of breast cancer survivors with lymphedema.

ELIGIBILITY:
Inclusion Criteria:

1. have a history of breast cancer;
2. previous diagnosis of lymphedema;
3. Stage II lymphedema based upon International Society of Lymphedema (the limb is firm in places, elevation does not reduce swelling, it may or may not pit with pressure, and skin changes may be noted);
4. be age 18 or older;
5. be able to see and read printed documents in English; and for stage 2 only,
6. have access to the Internet or a smart phone.

Exclusion Criteria: will not be:

1. undergoing chemotherapy or radiation, or
2. receiving hospice care. Additional exclusion criteria for local participants undergoing bioelectrical impedance measurements: pregnancy, metal implants, and defibrillator implants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2013-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
symptom burden | change between baseline and 1, 3, 6, and 12 months post-intervention
  self-report of symptoms will be documented on study instruments
function | change between baseline and 1, 3, 6, and 12 months post-intervention
  Self-report functional data using a validated instrument
psychological well-being | change between baseline and 1, 3, 6, and 12 months post-intervention
  self-report using a validated instrument

SECONDARY OUTCOMES:
coping | change between baseline and 1, 3, 6, and 12 months post-intervention
  self-report using validated instrument
self-care activities | Change between baseline 1, 3, 6, and 12 months post-intervention
  self report using a self-care checklist
stress | change between baseline and 1, 3, 6, and 12 months post-intervention
  self-report using a validated instrument
self-efficacy | change between baseline and 1, 3, 6, and 12 months post-intervention
  self-report using a validated instrument
social support | change between baseline and 1, 3, 6, and 12 months post-intervention
  self-report using a validated instrument
extracellular fluid | change between baseline and 3, 6, and 12 months post-intervention
  bioelectrical impedence measurement for sub set of participants

CONTACTS AND LOCATIONS:
Overall Officials: sheila h ridner, Phd, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt Univeristy School of Nursing, Nashville, Tennessee, United States